CLINICAL TRIAL: NCT06445595
Title: Investigation of the Effectiveness of Obesity in the Development of Chronic Headache After Traumatic Brain Injury
Brief Title: The Relationship Between Obesity and Chronic Headache
Status: Recruiting | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, HATİCE TOPRAK, asst. prof, Karaman Training and Research Hospital
Other Study IDs: 05-2024/19
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patients with traumatic brain injury — Patients will be contacted by phone
  Other Names: Patients will be contacted by phone

SUMMARY:
The relationship between obesity and the development of chronic headache after traumatic brain injury will be investigated.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) can be defined as an injury caused by an external force, particularly a direct blow to the head or exposure to a shock wave. In addition to the well-known consequences of TBI, including cognitive changes, motor deficits and sensory abnormalities, available evidence suggests that acute and chronic pain is also common after TBI. Obesity and TBI can be considered as public health problems with their increasing prevalence in recent years. Chronic pain adds to the already enormous clinical, psychological, social and economic burden of obesity. Developing mechanisms to prevent the development of pain after TBI has attracted the attention of researchers. Obesity is a preventable and modifiable clinical condition. The extent to which obesity may create adverse conditions after TBI remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 who suffered a head injury

Exclusion Criteria:

* People with severe head trauma
* Those who do not speak Turkish
* Those with a history of chronic opioid user
* Those with alcohol and drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals over the age of 18 who suffered a head injury
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The relationship between Bady Mass Index (BMI) and the development of chronic headache | Postoperative 3 month.
  BMI is calculated by dividing weight in kilograms by the square of height in metres.

SECONDARY OUTCOMES:
The relationship between the nature of trauma and the development of chronic headache | Postoperative 3 month.
  Head traumas that occur due to different reasons will be examined
The relationship between patients' education levels and chronic headache | Postoperative 3 month
  Education levels will be defined as primary school, secondary school and university graduate.

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Sharing will be evaluated in cases where the responsible researcher is contacted.